CLINICAL TRIAL: NCT07295262
Title: ICG-Cisplatin Self-Assembled Nanoprobes for Near-Infrared-Il Fluorescence Imaging-Guided Liver Resection
Brief Title: NIR-II Fluorescence-Guided Hepatectomy Using ICG-Cisplatin Nanoprobes for HCC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Jiwei Huang, Clinical Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JHuang20233
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Liver Cancer, Adult
Keywords: liver cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: NIR-II NanoM Group (Experimental): Patients receive transarterial embolization (TAE) with ICG-Cisplatin self-assembled nanoprobes (NIR-II NanoM) mixed with lipiodol, followed by fluorescence-guided laparoscopic anatomic hepatectomy.
  Interventions: Drug: ICG-Cisplatin Nanoprobe (NIR-II NanoM); Procedure: Fluorescence-guided Hepatectomy

INTERVENTIONS:
Drug: ICG-Cisplatin Nanoprobe (NIR-II NanoM) — Self-assembled nanoprobes of Indocyanine Green (ICG) and Cisplatin mixed with lipiodol (Shift&NanICG), administered via superselective transarterial injection for tumor staining.
Procedure: Fluorescence-guided Hepatectomy — Laparoscopic anatomic hepatectomy guided by Near-Infrared II (NIR-II) fluorescence imaging system to visualize tumor boundaries.

SUMMARY:
This prospective, single-arm exploratory study evaluates the feasibility and safety of a novel ICG-Cisplatin self-assembled nanoprobe (NIR-II NanoM) for fluorescence-guided surgery in patients with Hepatocellular Carcinoma (HCC). Participants will receive a transarterial injection of the nanoprobe mixed with lipiodol prior to surgery. During the subsequent laparoscopic anatomic hepatectomy, surgeons will utilize a Near-Infrared II (NIR-II) imaging system to visualize tumor boundaries and liver segments for precise resection.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years.
2. First diagnosis of Hepatocellular Carcinoma (HCC) (non-recurrent).
3. Single tumor with diameter ≤ 5 cm.
4. Assessed as resectable by more than 2 senior liver surgeons (experience >10 years, >500 hepatectomies).
5. No distant metastasis on preoperative chest CT and abdominal contrast-enhanced CT.
6. Child-Pugh Class A liver function.
7. Patient or legal guardian able to understand the study and sign informed consent.

Exclusion Criteria:

1. Postoperative pathology confirms cholangiocarcinoma, sarcomatoid HCC, combined HCC-ICC, or fibrolamellar carcinoma.
2. Presence of portal vein, hepatic vein, or bile duct tumor thrombus.
3. History of other malignancies (except cured carcinoma in situ of cervix, basal cell carcinoma, or squamous cell skin carcinoma).
4. Evidence of residual lesion, recurrence, or metastasis during preoperative assessment; or postoperative pathology confirming lymph node metastasis or positive margins.
5. Moderate to severe ascites requiring therapeutic paracentesis/drainage, or Child-Pugh score > 7 (except for small amount of ascites on imaging without clinical symptoms).
6. Uncontrolled or moderate/large amount of pleural effusion or pericardial effusion.
7. Severe cardiac, pulmonary, or renal dysfunction.
8. Ruptured HCC requiring emergency surgery.
9. Patient or family unable to understand the study conditions and objectives.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
3-Year Recurrence-Free Survival (RFS) | Up to 3 years post-surgery
  Calculated from the date of surgery to the date of first documented recurrence (local or distant) or death from any cause.
Rate of Successful Fluorescence Staining | Intraoperative (Day 0)
  The proportion of participants with successful visualization of the tumor. Success is defined as the NIR-II nanoprobe showing clear fluorescence signals in the tumor tissue under the NIR-II imaging system during surgery, enabling the surgeon to distinguish tumor boundaries and liver segments for precise resection.

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of surgery up to 3-5 years
  OS is defined as the time interval from the date of surgical resection to the date of death from any cause. For participants who are lost to follow-up, the last known contact date will be used as the censorship time.
Incidence of Perioperative Adverse Events and Complications | From enrollment through 30 days post-surgery
  The number of participants experiencing adverse events related to the nanoprobe (e.g., allergic reactions, nephrotoxicity) or surgical complications (e.g., bleeding, infection, bile leakage, liver failure). Events will be monitored and recorded according to standard clinical practice.
Rate of Local Recurrence | From date of surgery up to 3 years
  The percentage of participants who develop tumor recurrence specifically in the original surgical area (resection margin or tumor bed), with or without an elevation in tumor markers.
Rate of Distant Metastasis | From date of surgery up to 3 years
  The percentage of participants with metastasis detected in distant organs (e.g., lung, bone) or other liver segments. Metastasis is confirmed by CT, MRI, or nuclear scan without the mandatory need for pathological biopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No